CLINICAL TRIAL: NCT00365586
Title: A Phase III Study of the Efficacy, Tolerability and Safety of the Ketoprofen Topical Patch, 20% (KTP) in the Treatment of Pain Associated With Osteoarthritis Flare of the Knee, Including a Randomized, Double-Blind, Placebo-Controlled, Parallel Group Phase Followed by an Open-Label Treatment Phase
Brief Title: Ketoprofen Topical Patch, 20% in the Treatment of Pain Associated With Osteoarthritis Flare of the Knee
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: APR Applied Pharma Research s.a. (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: EN3269-303
Record Dates: First submitted 2006-08-16; First posted 2006-08-17 (Estimated); Last update posted 2020-02-19 (Actual); Status verified 2020-02

CONDITIONS: Osteoarthritis
Keywords: Pain; Osteoarthritis; Knee; NSAID
MeSH Terms: conditions — Osteoarthritis; Pain

INTERVENTIONS:
Drug: Ketoprofen Topical Patch , 20%

SUMMARY:
The purpose of this study is to evaluate the effect of a ketoprofen topical patch on the pain associated with Osteoarthritis Flare of the Knee.

DETAILED DESCRIPTION:
This randomized, double-blind placebo-controlled parallel group study will be conducted with patients who have experienced a flare of osteoarthritis of the knee. At screening, patients whose pain is currently controlled by an analgesic will agree, after giving Informed Consent, to discontinue that analgesic. Eligible patients will be randomized (1:1 ratio) to receive double-blind treatment with either the ketoprofen topical patch or a matching placebo patch to be applied once daily for 28 days. Patients will return to the clinic on Days 7, 14, 21 and 28. At Day 28, patients may choose to open a 2 month open-label period.

Patients will rate their pain using the Knee Injury and Osteoarthritis Outcome Score (KOOS) which contains the WOMAC pain subscale. Patients will also complete an electronic diary in which pain intensity, pain relief, and quality of sleep ratings will be captured. In addition, rescue medication consumption data will be collected. Ibuprofen will be provided as prn rescue medication.

ELIGIBILITY:
Inclusion Criteria:

* Males or females 18 years of age or older
* Diagnosis of osteoarthritis of the knee (unilateral or bilateral)
* Meet pain entry criteria
* Willing to discontinue use of all analgesic medications (including over-the-counter [OTC] analgesics) except those provided as the study treatment and rescue medication specifically for study purposes.

Exclusion Criteria:

* Positive urine pregnancy test, pregnant or lactating.
* Have fibromyalgia, inflammatory arthritis, gout, pseudo-gout or Paget's disease
* Have any other type of clinically significant joint disease or have had joint replacement surgery at the index knee
* Have received either a corticosteroid injection in the 4 weeks preceding the screening visit or hyaluronic acid within 6 months of the screening visit
* Have a history or physical examination finding that is incompatible with safe participation in the study or study product use
* Are taking medications or other substances contraindicated due to the nature of the study medication or the potential for drug interactions.
* Have significant renal or hepatic impairment
* Are taking a sleep medication at a dose that has not been stable for at least 3 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2006-08; Primary Completion 2007-04 (Actual); Study Completion 2007-05 (Actual)

PRIMARY OUTCOMES:
Pain as measured by the pain subscale of the Western Ontario and McMaster Universities (WOMAC) Osteoarthritis Index at Week 2

SECONDARY OUTCOMES:
Pain intensity, pain relief (diary)
Functional disability
Use of prn rescue medication
Quality of sleep
Lost days of work
Patient's and physician's global assessments of study medication

CONTACTS AND LOCATIONS:
Overall Officials: PPD, Principal Investigator — PPD Development, LP
Locations (1):
- PPD, Austin, Texas, United States